CLINICAL TRIAL: NCT01000246
Title: Response to Influenza Virus Vaccination in Patients Immunocompromised Due to Chemotherapy
Acronym: RIFLUVAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: O. de Weerdt, internist, Sint Antonius Hospital Nieuwegein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RIFLUVAC; version 2, 21-08-09
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Mamma Carcinoma; Heart Failure
Keywords: mammacarcinoma; breastcancer; chemotherapy; heart failure; influenza virus vaccine
MeSH Terms: conditions — Heart Failure; Influenza, Human | interventions — Influenza Vaccines; influvac; vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- influenza vaccine day 4 (Experimental): influenza vaccine day 4 of chemotherapy
  Interventions: Biological: influenza virus vaccine (influvac or vaxigrip)
- influenza vaccine day 16 (Experimental): influenza vaccine day 16 of chemotherapy
  Interventions: Biological: influenza virus vaccine (influvac or vaxigrip)
- influenza vaccine (Active Comparator): influenza vaccine in patients with heartfailure
  Interventions: Biological: influenza virus vaccine (influvac or vaxigrip)

INTERVENTIONS:
Biological: influenza virus vaccine (influvac or vaxigrip) — one i.m. dose of 0.5 mL
  Other Names: Influvac, MA number RVG 22289, ATC code J07BB02; Vaxigrip, MA number RVG 22306, ATC code J07BB02

SUMMARY:
Patients treated with chemotherapy or immunosuppressives are at higher risk of influenza infection and mortality and morbidity are higher compared to healthy adults. Vaccination against the influenza virus can prevent these complications. In this study it is investigated whether vaccination during chemotherapy is effective in reaching protective serum antibody concentrations and the relation between time of vaccination (day 4 +/- 1 day versus day 16 +/- 1 day of the chemotherapy cycle).

DETAILED DESCRIPTION:
This study will be conducted to answer the question whether vaccination during chemotherapy induces an adequate antibody response in oncology patients. Moreover, the effect of the timing of the vaccination during a chemotherapy cycle will be evaluated. In the mamma carcinoma patients, the effect of early versus late vaccination during a chemotherapy cycle will be studied. It was chosen to vaccinate in the early group at day 4 +/- 1 day; the immediate influence of the chemotherapy on the vaccination response is expected to have passed by then and patients will not already have their nadir. Late vaccination was defined as vaccination on day 16 +/- 1 day of the cycle. It is expected that the white blood cell and platelet counts by then are normalised.

In order to define a relatively homogenous patient population with mamma carcinoma, in this study patients will be recruited who are treated in the adjuvant setting with FEC-containing regimens (5-fluorouracil 500 mg/m2, epirubicin 100 mg/m2 and cyclophosphamid 500 mg/m2). The results of vaccination in these immunocompromised groups will be compared to the serological response to vaccination in persons who receive the influenza vaccination due to heart failure. Studies have shown that, although cytotoxic T-cell responses might be diminished, the rise in haemagglutinin inhibition titres in patients with heart failure vaccinated against influenza can be compared to the response to vaccination in otherwise healthy persons. These patients with heart failure will therefore be used as a control group. Patients with heart failure who are on treatment with immunosuppressives like prednisolone will not be included, because prednisolone diminishes the response to vaccination. The heart failure patients will be vaccinated according to the standard influenza vaccination protocol in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mamma carcinoma treated with FEC-containing triweekly chemotherapy at moment of vaccination
* Patients with heart failure and therefore having an indication for the influenza vaccination
* Age ≥ 18 years
* Signing of informed consent

Exclusion Criteria:

* Fever at time of vaccination defined as a temperature of ≥ 38.5 °C.
* Previous/known allergic reaction to any of the components of the vaccines given, for example hypersensitivity to egg protein
* Thrombocytopenia (defined as < 50 * 109/L ) at moment of vaccination
* Treatment with prednisolone on moment of vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Adequate rise in antibody titre | three weeks

SECONDARY OUTCOMES:
Antibody titres against the influenza virus before and after vaccination | three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Okke de Weerdt, Drs, Principal Investigator — Sint Antonius Hospital Nieuwegein; Douwe Biesma, Prof, Dr, Study Director — UMC Utrecht
Locations (8):
- Netherlands (8):
  - Maxima Medisch Centrum, Eindhoven, North Brabant
  - Medisch Centrum Alkmaar, Alkmaar, North Holland
  - Spaarne Ziekenhuis, Hoofddorp, North Holland
  - Martini Hospital Groningen, Groningen, Provincie Groningen
  - Maasstadziekenhuis, Rotterdam, South Holland
  - Meander Medisch Centrum, Amersfoort, Utrecht
  - Tergooiziekenhuizen, Blaricum, Utrecht
  - Sint Antonius Hospital, Nieuwegein, Utrecht